CLINICAL TRIAL: NCT03572192
Title: Tissue Collection Framework To Improve Outcomes In Solid Tumours
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 9094QM
Record Dates: First submitted 2018-06-18; First posted 2018-06-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumours

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background:

Cancer therapies have significantly improved over the last decades, allowing cancer specialists to keep cancer under control for longer than ever before. However, metastatic cancer still develops in a large number of patients and drug resistance occurs in the majority of them after an initial period of response and leads to cancer progression and death.

Aims:

To date, the mechanisms which allow cancer cells to spread through the body to form metastases and to become resistant even to the most powerful treatments are poorly understood. Our aim is to collect cancer specimens and normal tissue specimens such as blood from patients with solid tumours and to analyse these samples with some of the latest molecular profiling technologies in the research laboratory. This comprehensive analysis should reveal what molecular defects fuel the growth of cancer cells adn what allows them to spread through the body and then develop resistance to cancer therapies. Such insights could subsequently lead to the development of better more improved treatments which prevent drug resistance, to novel molecular tests which can also predict which treatment is most likely to be effective and tolerable in individual patients.

Methods:

To achieve this, we aim to collect multiple samples from consenting patients starting from the diagnosis of a tumour to the time drug resistance develops more. Importantly, this study will collect tissues from interventional procedures which are performed as part of routine patient management of patients seen at Barts Health NHS trust. We will then apply molecular tests such as proteomics and DNA sequencing to these samples. Tissues which are left over after these tests have been applied will be stored in a licensed tissue bank to allow future research with novel technologies.

DETAILED DESCRIPTION:
Approximately 320,000 patients are diagnosed with some form cancer in the UK each year. Despite improved therapies, half of these patients still die of their disease, usually after the failure of anticancer drug treatment. To date, mechanisms of drug resistance and also determinants of treatment toxicity which varies significantly between individual patients are poorly understood. Recent advances in molecular profiling techniques allow the comprehensive interrogation of large numbers of genes, transcripts and proteins which may be altered and contribute to progression and drug resistance in tumour tissues.

These technologies, including genome wide RNA expression and methylation profiling and DNA sequencing can be used to analyse the causes of cancer drug resistance in detail and this information can subsequently be used to develop better cancer drugs which prevent or overcome resistance and prolong patient survival. Furthermore, molecular studies can help to understand why some patients develop excessive toxicities during treatment with drugs which are well tolerated by most patients. This could help to develop tests that predict which individual patients will not tolerate a specific drug.

Importantly, we recently demonstrated that individual human tumours can contain highly heterogeneous cancer cell populations, for example good and poor prognosis cancer cells within the same tumour. This intratumour heterogeneity may have hampered the identification of markers of drug sensitivity or tumour aggressiveness in the past as single tumour biopsies are unlikely to reveal this complexity. Thus, our project uses our established sample collection protocols to comprehensively sample surgical specimens. This will allow the analysis of intratumour heterogeneity and its impact on outcome which is an urgent clinical need.

Tumour tissues can also change their molecular characteristics over time, for example during treatment, which mandates the longitudinal collection of tissue and blood specimens in order to understand how treatment resistance develops. We and others have recently shown that blood samples can be used to obtain information about tumour progression without the need for rebiopsies (Gerlinger, unpublished results and Forshew et al. Sci Transl Med 2012, 4:136ra68). Our aim is to regularly collect blood specimens from which tumour DNA and tumour cells can be extracted and studies as a surrogate of the tumour lesions. Taken together, multiregion sampling of tumours at surgery and longitudinal monitoring of molecular alterations over time should provide crucial insights into tumour heterogeneity and tumour evolution critical for progression and drug resistance.

The understanding of mechanisms of tumour progression also requires the use of cancer model systems in the laboratory and established cancer cell lines are generally used for this purpose. Such cell lines have often adapted to the laboratory tissue culture environment which changed their characteristics over time. Thus, they frequently behave differently from cells isolated directly from fresh tumour specimens, hindering their use for the identification of drug targets and resistance mechanisms. To circumvent this limitation, we will also use the collected tissues to isolate primary tumour and stromal cells and to maintain them in the laboratory for a limited period of time. This will provide the opportunity to study tumour characteristics in greater detail and will prevent false conclusions which can arise from artifacts which cannot be avoided in long term tissue culture.

Together, these efforts should improve our understanding of tumour evolution over time and reveal some of the mechanisms whih allow tumours to spread through the body and to develop cancer drug resistance. This will be a major improvement over traditional approaches which have most likely failed to identify mechanisms of cancer progression and treatment failure because they relied on single biopsies, missing heterogeneous changes in individual tumours and changes occurring over time (for further information: see Gerlinger et al (NEJM, March 2012) and Yap et al (Sci Transl Med, March 2012).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients over the age of 18 years who have been diagnosed with a solid tumour and who are seen at the Barts Health NHS Trust for clinical management of their tumour.
2. Male or female more than 18 years of age
3. Able to participate in the study.
4. Able to give informed consent.
5. Patients enrolled into other clinical trials may be included into this study

Exclusion Criteria

1. Any co-existing medical condition that in the Investigator's judgement will substantially increase the risk associated with the patient's participation in the study
2. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary studies
3. Physical or mental health issues that preclude them from participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: solid tumours
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2013-09; Primary Completion 2043-08 (Estimated); Study Completion 2043-08 (Estimated)

PRIMARY OUTCOMES:
Identification of molecular determinants of drug resistance, tumour progression or treatment toxicity. | 30years

CONTACTS AND LOCATIONS:
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom